CLINICAL TRIAL: NCT04925986
Title: Phase 2 Trial of Sitravatinib Plus Pembrolizumab in Patients With Advanced Treatment-Naïve PD-L1+ Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Sitravatinib Plus Pembrolizumab in Patients With Advanced Treatment-Naïve PD-L1+ Non-Squamous NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on data from other clinical trials
Sponsor: Sarah Goldberg (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sarah Goldberg, Associate Professor of Internal Medicine (Medical Oncology), Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000030093
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Diseases; Lung Neoplasms; Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7; PD-L1 Gene Mutation; Advanced Treatment-Naïve PD-L1; Sitravatinib; Pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases; Lung Neoplasms | interventions — sitravatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1A: PD-L1 1-49%, Main Study Population (Experimental): Participants with PD-L1 Tumor Proportion Score (TPS) 1-49% receive Pembrolizumab 200mg intravenous (IV) every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily, beginning on cycle 1 day 1 (C1D1).
  Interventions: Drug: Sitravatinib; Drug: Pembrolizumab
- Group 1B: PD-L1 1-49%, Pembrolizumab run-in population (Experimental): Participants with PD-L1 Tumor Proportion Score (TPS) 1-49% receive Pembrolizumab 200mg intravenous (IV) for one dose alone, beginning on cycle 1 day 1 (C1D1). On Cycle 2 Day 1 (C2D1), participants receive Pembrolizumab 200mg intravenous (IV) once every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily.
  Interventions: Drug: Sitravatinib; Drug: Pembrolizumab
- Group 2A: PD-L1 ≥ 50%, Main Study Population (Experimental): Participants with PD-L1 Tumor Proportion Score (TPS) ≥ 50% receive Pembrolizumab 200mg intravenous (IV) every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily, beginning on cycle 1 day 1 (C1D1).
  Interventions: Drug: Sitravatinib; Drug: Pembrolizumab
- Group 2B: PD-L1 ≥ 50%, Pembrolizumab run-in population (Experimental): Participants with PD-L1 Tumor Proportion Score (TPS) ≥ 50% receive Pembrolizumab 200mg intravenous (IV) for one dose alone, beginning on cycle 1 day 1 (C1D1). On Cycle 2 Day 1 (C2D1), participants receive Pembrolizumab 200mg intravenous (IV) once every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily.
  Interventions: Drug: Sitravatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sitravatinib — Groups 1A and 2A receive Sitravatinib 100mg orally (PO) daily starting on cycle 1 day 1 (C1D1). Groups 1B and 2B) receive Sitravatinib 100mg orally (PO) daily starting on Cycle 2 Day 1 (C2D1).
  Other Names: IND 155305
Drug: Pembrolizumab — All groups (1A, 1B, 2A, 2B) receive Pembrolizumab 200mg intravenous every three weeks (IV Q3w) on cycle 1 day 1 (C1D1).
  Other Names: Keytruda

SUMMARY:
This is a multicohort phase 2 study to evaluate the efficacy of pembrolizumab combined with the investigational drug sitravatinib in the frontline treatment of advanced, non-squamous PD-L1 positive NSCLC.

DETAILED DESCRIPTION:
This is a multicohort phase 2 study to evaluate the efficacy of pembrolizumab combined with the investigational drug sitravatinib in the frontline treatment of advanced, non-squamous PD-L1 positive NSCLC. For clinical analysis, there will be two patient cohorts defined by PD-L1 status: Cohort 1 for patients with PD-L1 Tumor Proportion Score (TPS) 1-49% and Cohort 2 for patients with TPS≥50%. The investigators will implement a Simon's two-stage design to evaluate the efficacy of sitravatinib in combination with pembrolizumab for each cohort separately.

There will be two groups within each cohort of this study: the "main study population" (Group A) in which patients will receive pembrolizumab plus sitravatinib beginning on Cycle 1 Day 1 (C1D1), and a "pembrolizumab run-in population" (Group B) in which patients will receive pembrolizumab alone for 1 dose followed by pembrolizumab plus sitravatinib beginning C2D1.

The primary endpoint of the trial is the ORR for patients treated with pembrolizumab plus sitravatinib in the main study population. The purpose of the pembrolizumab run-in population is to obtain tissue and blood samples from these patients to be used as controls for correlative studies and to determine the preliminary efficacy of pembrolizumab alone followed by the combination.

Primary Objective

(1) The primary objective of this study is to evaluate the efficacy of sitravatinib in combination with pembrolizumab in the front-line treatment of patients with advanced non-squamous PD-L1 positive NSCLC by measuring Objective Response Rate (ORR).

Secondary Objectives

1. To evaluate other measures of efficacy including Overall Survival (OS), Progression Free Survival (PFS), Duration of Response (DOR) and Clinical Benefit Rate (CBR) in the first-line setting for patients with advanced, non-squamous, PD-L1 positive NSCLC treated with the combination of sitravatinib and pembrolizumab.
2. To evaluate the toxicity profile and tolerability of sitravatinib/pembrolizumab in advanced, treatment naïve, non-squamous, PD-L1 positive NSCLC.

Exploratory Objectives:

1. To evaluate ORR, OS, PFS, DOR, and CBR in patients with advanced, non-squamous, treatment naïve, PD-L1 positive NSCLC who receive pembrolizumab run-in followed by pembrolizumab/sitravatinib combination therapy.
2. To evaluate the CNS activity of sitravatinib/pembrolizumab in patients with advanced, treatment naïve, PD-L1 positive NSCLC by measuring Intracranial Objective Response Rate (iORR) and Intracranial Duration of Response(iDOR) in patients with baseline CNS disease, and Intercranial Progression-Free Survival (iPFS) in all patients.
3. To study correlates of the adaptive and innate immune responses induced by sitravatinib and pembrolizumab treatment in both tumor tissue and peripheral blood.
4. To explore the association between tumor immune contexture and clinical benefit to sitravatinib and pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

In order to be to be eligible to participate in this study, an individual must meet all of the following criteria:

* Histologically or cytologically confirmed non-squamous NSCLC that is metastatic (Stage IV), recurrent, or unresectable locally advanced (Stage IIIB/IIIC) disease, not amenable to treatment with curative intent.
* No prior systemic therapy for advanced disease. Prior chemotherapy for local or locally advanced disease is allowed if completed >6 months prior to trial enrollment. Prior immunotherapy is not allowed.
* PD-L1 ≥ 1% using the 22c3 PD-L1 IHC assay or a local assay performed in a CLIA facility
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Life expectancy of at least 3 months.
* Measurable disease as per RECIST v1.1
* Adequate bone marrow and organ function demonstrated by:

  * Absolute neutrophil count >1,500/mm3 (1.5 × 10^9/L).
  * Hemoglobin ≥ 8.0 g/dL not dependent on transfusion support.
  * Platelet count ≥ 75 × 10^9/L (≥ 75,000 per mm3).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN without liver metastases; < 5.0 x ULN if documented liver metastases
  * Serum total bilirubin ≤ ULN, or for patients with potential Gilbert's, direct bilirubin ≤ ULN
  * Calculated creatinine clearance ≥ 40 mL/min, using the Cockcroft-Gault formula.
* Women of child-bearing potential (WOCBP) or men whose partner is a WOCBP agrees to use contraception while participating in this study, and for a period of 6 months following termination of study treatment.
* Completed informed consent process, including signing IRB approved informed consent form.
* Willing to comply with clinical trial instructions and requirements.
* Willing to undergo an on-treatment biopsy with an appropriate biopsy site identified prior to treatment initiation

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Symptomatic or untreated brain metastases ≥ 2cm in diameter. Patients with brain lesions that are adequately treated with local therapy (i.e. radiation therapy) and neurologically stable without the need for corticosteroids for at least 2 weeks prior to enrollment are allowed. Patients with brain lesions that are asymptomatic, smaller than 2cm, in non-critical regions of the brain and not requiring corticosteroids for at least 2 weeks prior to enrollment may be eligible after review with the Sponsor Investigator.
* Leptomeningeal disease
* Known mutations/alterations in EGFR, ROS1, ALK, or BRAF
* Any prior treatment with checkpoint inhibitor therapy or other immunotherapy agents
* Any prior treatment with therapy having the same mechanism of action as sitravatinib (e.g., tyrosine kinase inhibitor with a similar target profile or bevacizumab/ramucirumab)
* Active or prior documented autoimmune disease within the past 2 years (note: patients with type 1 diabetes, vitiligo, Graves' disease, hypothyroidism due to an autoimmune condition only requiring hormone replacement, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded).
* Active or prior immunocompromising conditions, including use of immunosuppressive medication within 2 weeks of enrollment. This does not include topical, intranasal or inhaled steroids with minimal systemic absorption or systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or equivalent. Use of higher dose corticosteroids for short/defined course (ie prophylaxis in patients with contrast dye allergy) is also allowed if indicated.
* Uncontrolled HIV. Patients with HIV may be eligible if they meet the following criteria:

  * CD4+ T cell count>350 cell/uL
  * No history of AIDS-defining opportunistic infection within the past 12 months
  * Currently tolerating treatment with ART for at least 4 weeks prior to enrollment, with HIV viral load <400 copies/mL
  * Patients on specific ART drugs with possibility for drug-drug interaction with sitravatinib may be excluded (see appendix 5).
* Active hepatitis C (HCV) infection. Patients with a history of HCV may be eligible if they have completed curative antiviral treatment with undetectable HCV viral load and liver function tests are otherwise within acceptable limits (as described in Section 4.5.2). Patients with chronic Hepatitis B (HBV) infection are not excluded if liver function is within acceptable limits, but should be evaluated for reactivation risk and started on suppressive antiviral therapy prior to enrollment if appropriate.
* History of stroke or transient ischemic attack within the previous 6 months.
* History of life threatening venous thromboembolic event (such as hemodynamically significant pulmonary embolism) or any arterial thrombotic event within the previous 6 months. Patients with non-life threatening venous thromboembolic events are not excluded and should be managed with anti-coagulation as per standard institutional practice.
* Any of the following cardiac abnormalities:

  * Unstable angina pectoris within the past 6 months.
  * Congestive heart failure ≥ NYHA Class 3 within the past 6 months.
  * Prolonged QTc on electrocardiogram >500 milliseconds.
  * Left ventricular ejection fraction (LVEF) < 40%.
* Uncontrolled hypertension (>150mm Hg or >100mm Hg diastolic) on multiple observations despite standard of care treatment
* Major surgery within 4 weeks of the date of randomization.
* History of significant hemoptysis or hemorrhage within 4 weeks of the date of randomization.
* Known or suspected presence of another malignancy that could be mistaken for the malignancy under study during disease assessments.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Pregnancy. WOCBP must have a negative serum or urine pregnancy test documented within the screening period prior to the date of randomization.
* Breast-feeding or planning to breast-feed during the study or within 30 days following the last dose of sitravatinib and within 5 months following the last dose of pembrolizumab.
* Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Goldberg, MD MPH, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1A: PD-L1 1-49%, Main Study Population | Group 1B: PD-L1 1-49%, Pembrolizumab run-in Population | Group 2A: PD-L1 ≥ 50%, Main Study Population | Group 2B: PD-L1 ≥ 50%, Pembrolizumab run-in Population
Started | 1 | 2 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 3 | 3
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sitravatinib: Group 1A; Sitravatinib: Group 2A: Participants receive Pembrolizumab 200mg intravenous (IV) every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily, beginning on cycle 1 day 1 (C1D1).
  Sitravatinib: Groups 1A and 2A receive Sitravatinib 100mg orally (PO) daily starting on cycle 1 day 1 (C1D1). Groups 1B and 2B) receive Sitravatinib 100mg orally (PO) daily starting on Cycle 2 Day 1 (C2D1).
  Pembrolizumab: All groups (1A, 1B, 2A, 2B) receive Pembrolizumab 200mg intravenous every three weeks (IV Q3w) on cycle 1 day 1 (C1D1).
- Sitravatinib Group 1B; Sitravatinib Group 2B: Participants with receive Pembrolizumab 200mg intravenous (IV) for one dose alone, beginning on cycle 1 day 1 (C1D1). On Cycle 2 Day 1 (C2D1), participants receive Pembrolizumab 200mg intravenous (IV) once every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily.
  Sitravatinib: Groups 1A and 2A receive Sitravatinib 100mg orally (PO) daily starting on cycle 1 day 1 (C1D1). Groups 1B and 2B) receive Sitravatinib 100mg orally (PO) daily starting on Cycle 2 Day 1 (C2D1).
  Pembrolizumab: All groups (1A, 1B, 2A, 2B) receive Pembrolizumab 200mg intravenous every three weeks (IV Q3w) on cycle 1 day 1 (C1D1).
- Total: Total of all reporting groups
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A | Sitravatinib Group 1B | Sitravatinib Group 2B | Total
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 0 | 3
  >=65 years | 0 | 2 | 1 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 5
  Male | 1 | 2 | 0 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 2 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 3 | 2 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 2 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The Objective Response Rate (ORR): The primary endpoint for this study will be ORR as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) in the main study population. Presented are counts of participants in the following RECIST categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD)
Time Frame: up to 267 days
Population: Participants available for assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Sitravatinib: Group 1B; Sitravatinib: Group 2B: Participants receive Pembrolizumab 200mg intravenous (IV) for one dose alone, beginning on cycle 1 day 1 (C1D1). On Cycle 2 Day 1 (C2D1), participants receive Pembrolizumab 200mg intravenous (IV) once every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily.
  Sitravatinib: Groups 1A and 2A receive Sitravatinib 100mg orally (PO) daily starting on cycle 1 day 1 (C1D1). Groups 1B and 2B) receive Sitravatinib 100mg orally (PO) daily starting on Cycle 2 Day 1 (C2D1).
  Pembrolizumab: All groups (1A, 1B, 2A, 2B) receive Pembrolizumab 200mg intravenous every three weeks (IV Q3w) on cycle 1 day 1 (C1D1).
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A | Sitravatinib: Group 1B | Sitravatinib: Group 2B
Number analyzed (Participants) | 1 | 2 | 2 | 3
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 1 | 1
  Stable Disease (SD) | 1 | 2 | 0 | 2
  Progressive Disease (PD) | 0 | 0 | 1 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) in the main study populations (ie groups 1A and 2A) is a secondary endpoint for this study. OS in groups 1B and 2B is an exploratory endpoint. Defined as the time from date of treatment start to death due to any cause
Time Frame: until death or date of last contact, up to 2 years
Population: Only patients who met the eligibility criteria were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A
Number analyzed (Participants) | 1 | 3
days | 246 [NA to NA] — Due to insufficient number of participants with events, confidence intervals could not be calculated. | 210 [24 to NA] — Due to insufficient number of participants with events, upper limit could not be calculated.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) in the main study populations (ie groups 1A and 2A) is a secondary endpoint for this study. PFS in groups 1B and 2B is an exploratory endpoint. Defined as time from first dose to first progressive disease (PD) or death due to any cause in the absence of documented PD.
Time Frame: Until progressive disease, death, or last contact, up to 2 years
Population: Only patients who met the eligibility criteria were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A
Number analyzed (Participants) | 1 | 3
days | 246 [NA to NA] — Due to insufficient number of participants with events, confidence intervals could not be calculated. | 210 [24 to NA] — Due to insufficient number of participants with events, upper limit could not be calculated.

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) for patients in Group A is a secondary endpoints for this study; DOR for Group B is an exploratory endpoint. Defined as time that measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or to death due to any cause in the absence of documented PD.
Time Frame: Until progressive disease, death, or last contact, up to 2 years
Population: Data for this outcome was not collected as there were no patients that met criteria for CR or PR.
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) in Group A is a secondary endpoints for this study, while CBR in Group B is an exploratory endpoint. Defined as percent of patients documented to have a confirmed Complete Response (CR), confirmed Partial Response (PR), or Stable Disease (SD) documented on at least 1 on-study assessment and including at least 5 weeks on study
Time Frame: up to 2 years
Population: Only patients who met the eligibility criteria were analyzed. For paricipants in Group 2A, 2 had confirmed SD and 1 was unevaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A
Number analyzed (Participants) | 1 | 3
percentage of participants | 100 | 66.7

6. Secondary Outcome: Number of Participants That Experienced at Least 1 Adverse Event
Description: Evaluation of the safety and toxicity profile of the combination of sitravatinib and pembrolizumab in the first-line treatment of patients with non-squamous metastatic NSCLC is a secondary objective in this study. Secondary endpoint is adverse events as per CTCAE v.5. The Safety population is defined as all patients who received any dose of study treatment (i.e., sitravatinib and/or pembrolizumab) and will be used for all safety analyses. Number of participants that experienced at least 1 adverse event.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A | Sitravatinib: Group 1B | Sitravatinib: Group 2B
Number analyzed (Participants) | 1 | 3 | 2 | 3
Participants | 1 | 3 | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to 450 days
Groups:
- Sitravatinib: Group 1A; Sitravatinib: Group 2A: Participants with PD-L1 Tumor Proportion Score (TPS) 1-49% receive Pembrolizumab 200mg intravenous (IV) every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily, beginning on cycle 1 day 1 (C1D1).
  Sitravatinib: Groups 1A and 2A receive Sitravatinib 100mg orally (PO) daily starting on cycle 1 day 1 (C1D1). Groups 1B and 2B) receive Sitravatinib 100mg orally (PO) daily starting on Cycle 2 Day 1 (C2D1).
  Pembrolizumab: All groups (1A, 1B, 2A, 2B) receive Pembrolizumab 200mg intravenous every three weeks (IV Q3w) on cycle 1 day 1 (C1D1).
- Sitravatinib: Group 1B; Sitravatinib: Group 2B: Participants with PD-L1 Tumor Proportion Score (TPS) 1-49% receive Pembrolizumab 200mg intravenous (IV) for one dose alone, beginning on cycle 1 day 1 (C1D1). On Cycle 2 Day 1 (C2D1), participants receive Pembrolizumab 200mg intravenous (IV) once every 3 weeks (Q3w) and Sitravatinib 100mg PO (by mouth) daily.
  Sitravatinib: Groups 1A and 2A receive Sitravatinib 100mg orally (PO) daily starting on cycle 1 day 1 (C1D1). Groups 1B and 2B) receive Sitravatinib 100mg orally (PO) daily starting on Cycle 2 Day 1 (C2D1).
  Pembrolizumab: All groups (1A, 1B, 2A, 2B) receive Pembrolizumab 200mg intravenous every three weeks (IV Q3w) on cycle 1 day 1 (C1D1).
Arm/Group | Sitravatinib: Group 1A | Sitravatinib: Group 2A | Sitravatinib: Group 1B | Sitravatinib: Group 2B
All-Cause Mortality (participants affected / at risk) | 1/1 | 2/3 | 2/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/3 | 2/2 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitravatinib: Group 1A (N=1) | Sitravatinib: Group 2A (N=3) | Sitravatinib: Group 1B (N=2) | Sitravatinib: Group 2B (N=3)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Subarachnoid bleeding (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitravatinib: Group 1A (N=1) | Sitravatinib: Group 2A (N=3) | Sitravatinib: Group 1B (N=2) | Sitravatinib: Group 2B (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 2
Double vision (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis, oral (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Edema of limbs (General disorders) | 0 | 0 | 1 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 2
Gait disturbance (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 2 | 1 | 0
Rash (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2
ALT increased (Investigations) | 0 | 1 | 1 | 2
AST increased (Investigations) | 0 | 1 | 1 | 2
Creatinine increased (Investigations) | 0 | 0 | 1 | 0
QTc prolongation (Investigations) | 1 | 0 | 0 | 0
Free T4 increased (Investigations) | 0 | 0 | 1 | 1
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 1
LDH increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Urine ketone elevated (Investigations) | 0 | 0 | 0 | 1
WBC elevated (Investigations) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 2 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid Bleeding (Nervous system disorders) | 0 | 0 | 1 | 0
Transient Ischemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Bactiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 1 | 2
Leukocytes in Urine (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopeica (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eyelashes Loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-Plantar Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Raynaud's Syndrome (Vascular disorders) | 0 | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT04925986/Prot_SAP_000.pdf